CLINICAL TRIAL: NCT07350434
Title: The Acute Effects of Neurodynamic Stretching on the Shear Wave Velocity: the Effects of Hip Adduction and Abduction
Brief Title: Hip Abduction and Adduction During Neurodynamic Stretching
Acronym: HIPROT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Burgundy (Other)
Responsible Party: Principal Investigator, Nicolas Babault, Prof, University of Burgundy
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CEP2601
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Stretching; Control Condition
Keywords: stretching; stiffness; nerve; muscle; flexibility; hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- No intervention (neutral) (No Intervention): No intervention with measurements in neutral position
- No intervention (adduction) (No Intervention): No intervention with measurements in adduction position
- No intervention (abduction) (No Intervention): No intervention with measurements in abduction position
- Neurodynamic (neutral) (Active Comparator): The hip was positioned neutral (alignment between the lower limb and the trunk).
  Interventions: Other: Maximal neurodynamic flossing
- Neurodynamic (adduction) (Experimental): The hip was positioned in adduction and the neurodynamic stretch was applied.
  Interventions: Other: Maximal neurodynamic flossing
- Neurodynamic (abduction) (Experimental): The hip was positioned in abduction and the neurodynamic stretch was applied.
  Interventions: Other: Maximal neurodynamic flossing

INTERVENTIONS:
Other: Maximal neurodynamic flossing — Neurodynamic flossing was applied at pain threshold on hamstring muscles and repeated 5 times during 60s at the point of pain. During the neurodynamic conditions, head and ankle movement permitted to mobilize nerve tissues. Flossing is the alternation of these movements every 2 seconds.
  Arms: Neurodynamic (abduction); Neurodynamic (adduction); Neurodynamic (neutral)

SUMMARY:
Neurodynamic mobilization techniques are widely applied in rehabilitation and physiotherapy to enhance the mobility and function of peripheral nerves. Two main approaches are distinguished : Nerve tensioning and nerve flossing. They both involve proximal and distal joint movements to induce greater neural sliding while avoiding excessive tensile stress. However, contradictory findings following neurodynamic stretching highlighted the current lack of consensus regarding the position that should be used. Moreover, neurodynamic techniques are of interest for patients, it appeared it could also be applied in healthy individuals and more particularly in athletes. Accordingly, the primary objective of the present study was to determine the immediate effect of two hip positions (adduction vs. abduction) during neurodynamic flossing techniques on the sciatic nerve and hamstring tissues using the shear wave elastography (SWE, a form of ultrasonography).

DETAILED DESCRIPTION:
Neurodynamic mobilization techniques are frequently applied in rehabilitation settings to enhance the mobility and function of peripheral nerves, particularly in the management of neuropathic pain such as carpal tunnel syndrome, radiculopathies, or sciatica. Two main approaches are distinguished. Nerve tensioning involves maintaining the nerve stretched at the end of the joint range of motion with relatively limited excursion. It is similar to a static stretching intervention but with distal (ankle) and proximal (cervical) tensions. Nerve flossing (also termed gliding or sliders), consists of alternating proximal and distal joint movements to induce greater neural sliding while avoiding excessive tensile stress. Both techniques appear efficient. However, contradictory findings following neurodynamic stretching highlighted the current lack of consensus regarding the angular position that could be used. For instance, hip rotations or hip adduction could impact muscle or nerve tissue changes, particularly in healthy tissues. Moreover, neurodynamic techniques are of interest for patients, it appeared it could also be applied in healthy individuals and more particularly in athletes. Performed in patients, healthy or athletes, no study has compared different hip positions. Accordingly, the primary objective of the present study was to determine the immediate effect of two hip positions (adduction vs. abduction) during neurodynamic flossing techniques on the sciatic nerve and hamstring tissues using the shear wave elastography (SWE, a form of ultrasonography). This method has been shown reliable to provide non-invasive real-time assessments of soft tissues elastic properties.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* physical active
* no injuries (lower limb or back pain) in the past 3 months

Exclusion Criteria:

* Specific lower limb (hamstring) injuries in the past 2 years
* Not restraining activity 24h before participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Nerve shear wave velocity using elastography in neutral position | Before the intervention and at the end (immediately after) the intervention
  Shear wave velocity of the sciatic nerve will be evaluated by using an ultrasound (echography) device with a specific mode called "shear wave elastography". Briefly, the ultrasound probe will deliver an ultrasound wave. The propagation speed (called '"shear wave velocity") will be measured by the same probe. The greater the velocity is, the harder the tissue is. The hip position was neutral (alignment between the lower limb and the trunk).

SECONDARY OUTCOMES:
Nerve shear wave velocity using elastography in experimental position | Before the intervention and at the end (immediately after) the intervention
  Shear wave velocity of the sciatic nerve will be evaluated by using an ultrasound (echography) device with a specific mode called "shear wave elastography". Briefly, the ultrasound probe will deliver an ultrasound wave. The propagation speed (called '"shear wave velocity") will be measured by the same probe. The greater the velocity is, the harder the tissue is. The hip position was the experimental position (i.e., adduction or abduction depending on the randomisation).
Muscle shear wave velocity using elastography in neutral position | Before the intervention and at the end (immediately after) the intervention
  Shear wave velocity of the biceps femoris muscle will be evaluated by using an ultrasound (echography) device with a specific mode called "shear wave elastography". Briefly, the ultrasound probe will deliver an ultrasound wave. The propagation speed (called '"shear wave velocity") will be measured by the same probe. The greater the velocity is, the harder the tissue is. The hip position was neutral (alignment between the lower limb and the trunk).
Muscle shear wave velocity using elastography in the experimental position | Before the intervention and at the end (immediately after) the intervention
  Shear wave velocity of the biceps femoris muscle will be evaluated by using an ultrasound (echography) device with a specific mode called "shear wave elastography". Briefly, the ultrasound probe will deliver an ultrasound wave. The propagation speed (called '"shear wave velocity") will be measured by the same probe. The greater the velocity is, the harder the tissue is. The hip position was the experimental position (i.e., adduction or abduction depending on the randomisation).
Hamstring force | Before the intervention and at the end (immediately after) the intervention
  Maximal torque during a maximal voluntary hamstring contraction
Biceps femoris electromyographic activity | Before the intervention and at the end (immediately after) the intervention
  Electromyographic activity of biceps femoris muscle
Semitendinosus electromyographic activity | Before the intervention and at the end (immediately after) the intervention
  Electromyographic activity of semitendinosus
passive knee extension | Before the intervention and at the end (immediately after) the intervention
  The final passive range of motion of the hamstring muscles
Global flexibility | Before the intervention and at the end (immediately after) the intervention
  the stand and reach test to evaluate flexibility (in centimeters)
Slump test | Before the intervention and at the end (immediately after) the intervention
  Seated flexibility using the slump test (in degrees)
discomfort | At the end (immediately after) the intervention
  rating of perceived discomfort during the intervention (from 1 to 10, no discomfort to maximal discomfort, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Babault, Principal Investigator — universite bourgogne europe
Locations (1):
- Universite Bourgogne Europe - faculty of sports sciences, Dijon, France

IPD SHARING:
Plan to Share IPD: Yes
data freely available in online websites